CLINICAL TRIAL: NCT04110080
Title: Enhanced Recovery After Surgery in Living Donor Kidney Transplant Donors
Brief Title: Enhanced Recovery After Surgery in Kidney Transplant Donors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19D.574
Record Dates: First submitted 2019-09-20; First posted 2019-10-01 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Opioid Use; Kidney Diseases; Pain, Postoperative; Postoperative Complications; Postoperative Nausea and Vomiting
Keywords: enhanced recovery after surgery; living donor kidney transplant; multimodal analgesia
MeSH Terms: conditions — Kidney Diseases; Pain, Postoperative; Postoperative Complications; Postoperative Nausea and Vomiting | interventions — Anesthesia, Conduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced recovery after surgery (Experimental): Preoperatively, patients will be counseled on optimization of physical and nutritional status. They will receive carbohydrate loading drinks prior to surgery. Intraoperatively, standard ASA monitors will be utilized, and patients will receive general anesthesia. Goal directed fluid management will be enforced with bolus options based on hemodynamics. Transabdominal plane and rectus sheath block will be performed in the operating room by the regional anesthesia team. Post-operatively pain management will include multimodal analgesic medications. Regular diet will be allowed and encouraged on post-operative day 0 (POD). Lines and drains will be minimized to encourage early mobilization and bowel function. Patients will be counseled on expectations of discharge criteria POD0.
  Interventions: Procedure: multimodal pain management; Other: goal directed fluid management; Other: preoperative carbohydrate loading; Procedure: Donor nephrectomy; Procedure: regional anesthesia
- Standard of care (Active Comparator): Patients will receive traditional care for donor nephrectomy. Patients will be instructed to fast for 24 hours preoperative. On day of surgery, standard monitors will be used, and intraoperative management per anesthesiologists discretion including pain management. Post-operative, patients will receive pain medications, including opioids, as needed. Intravenous fluids will be continued until patients tolerate liquids per os. Bowel regimen will be ordered as needed. Patients will be discharged once meeting pre-set criteria.
  Interventions: Procedure: Donor nephrectomy

INTERVENTIONS:
Procedure: multimodal pain management — Regional anesthesia techniques, specifically rectus sheath and transabdominal plane blocks, for pain management will be performed.
  Arms: Enhanced recovery after surgery
Other: goal directed fluid management — Intraoperatively fluids will be administered based on hemodynamic parameters, in addition to clinical judgement.
  Arms: Enhanced recovery after surgery
Other: preoperative carbohydrate loading — Patient's nutrition will be optimized preoperatively by administering carbohydrate drinks, and limiting fasting time.
  Arms: Enhanced recovery after surgery
Procedure: Donor nephrectomy — All patient will have laparoscopic nephrectomy procedure with transplant surgery.
Procedure: regional anesthesia — transabdominal plane and rectus sheath nerve block
  Arms: Enhanced recovery after surgery

SUMMARY:
Enhanced recovery after surgery (ERAS) pathways are designed to optimize perioperative management, improving patient outcomes and satisfaction through multimodal techniques. Living kidney transplant donors are typically healthy individuals who undergo laparoscopic nephrectomy. The most significant hindrance to discharge to return to activities of daily living is frequently return of bowel function and postoperative pain.

Through a randomized controlled trial design, we will evaluate the effectiveness of implementing an ERAS pathway. We hypothesize that preoperative patient optimization through exercise, carbohydrate loading, and counseling on expectations, in addition to multimodal pain management strategies which limit opioids would allow faster recovery, early bowel function, decreased postoperative pain, increased patient satisfaction and shorter length of stay.

The study population will include a total of 42 patients (age 18-80) who are American Society of Anesthesiologists (ASA) Physical Status (PS) 1-3, undergoing living donor nephrectomy. Our primary outcome measures will be postoperative opioid consumption. Secondary outcome measures are: postoperative pain score, time to return of bowel function, ambulation, first oral intake postoperatively, and patient satisfaction scores. Other objectives include reducing readmissions, shorter hospital length of stay and decreased operative complications, including nausea, vomiting and wound infection.

DETAILED DESCRIPTION:
ERAS pathways have been widely used in multiple surgical disciplines leading to improvements in perioperative care. The goal of the pathways is to decrease postoperative opioid consumption, improve pain scores, decrease length of hospital stay, lower morbidity, and increase patient satisfaction. Living kidney donors are in high demand and represent a large portion of grafts supplied for kidney transplant. The primary objective of our study is to initiate an enhanced recovery after surgery pathway designed to facilitate early recovery and to study the impact of an ERAS protocol on the living donor nephrectomy population.

The study is a prospective, randomized, controlled clinical trial evaluating the effect of ERAS to decrease postoperative opioid consumption, improve pain scores, decrease length of hospital stay, lower morbidity, and increase patient satisfaction. Patients will complete standard preoperative workup as per protocol for donor nephrectomy, and they will also be evaluated at the preadmission testing clinic. Consent will be obtained by a member of the research team at a preoperative office visit. At this time, patients will be randomized to enhanced recovery after surgery (ERAS) pathway or standard of care, and they will be informed on what to expect during their hospital course.

ERAS pathway:

Preoperatively, according to the ERAS pathway devised, patients will be counseled on optimization of physical status. They will be encouraged to sustain from smoking and alcohol, exercise daily, and encourage healthy diet. If the physician determines the need for nutritional counsel, they will have a workup by a nutritionist. They will also be labeled as ERAS pathway in the case request submitted by the surgeon. For the day of surgery, patients will receive carbohydrate drinks and dietary instructions. All patients will be instructed to have a clear liquid diet 24 hours prior to surgery with no food after midnight. Patients will receive 2 carbohydrate pre-surgery drinks (20 oz total) - 10oz for the night before surgery, and 10oz to drink within 1 hour of scheduled arrival time. On arrival the day of surgery, patients will receive the following medications, unless contraindicated or allergy: acetaminophen 1g PO, pregabalin 150 mg PO, and celecoxib 400 mg PO.

Patients will be evaluated in the preoperative holding area by a member of the anesthesiology staff. Peripheral IV will be placed. Patients will be screened for risk of post-operative nausea and vomiting (PONV) (female, nonsmoker, prior PONV, planned postoperative opioid each 1 point), if deemed high risk a scopolamine patch will be applied in holding. Patients will at that point be counseled on use of regional anesthesia for postoperative pain and additional consent for transabdominal plane and rectus sheath blocks will be obtained. Premedication with midazolam will be administered. Subcutaneous heparin 5000 units will be given prior to surgery, as per standard of care.

Intraoperatively, standard ASA monitors will be utilized, and patients will receive general anesthesia with propofol, fentanyl, rocuronium (dosed by weight), and sevoflurane maintenance for all patients. Additional IV access will be established. Antibiotics will be administered within 1 hour of incision per protocol. Goal directed fluid management with Plasmalyte or Lactated ringers with goal of 3-4 ml/kg/hr ideal body weight, with bolus option for clinical indications of MAP < 65mmHg. If requiring more than 2 boluses of 200-250 ml, phenylephrine infusion will be used for hypotension. Additional antiemetic prophylaxis will be given: ondansetron 4mg for all patients with the addition of dexamethasone 10 mg if high risk of PONV. At the end of the case, ketorolac 15 mg will be given.

The transabdominal plane and rectus sheath block will be performed in the operating room by the regional anesthesia team, after the skin is closed and dressings are applied but while the patient is still under general anesthesia. An ultrasound guided approach will be used to identify the plane between the internal oblique and transversus abdominis muscles. Twenty ml (10 ml each side) of 0.375% ropivacaine will be injected to anesthetize the nerves supplying the anterior abdominal wall (T6 to L1). For the rectus sheath block the ultrasound transducer will be positioned immediately lateral to umbilicus and 20 ml (10 ml each side) of 0.375% ropivacaine local anesthetic will be injected between rectus muscle and posterior rectus sheath.

Following extubation, patients will return to post-anesthesia care unit (PACU) and be discharged to their inpatient room per standard guidelines. Phenergan 6.25 mg IV BID or ondansetron 4mg IV q8 will be administered as needed for PONV. Additional pain management will includes ketorolac 15mg q6 for 48 hours post operatively, acetaminophen 1g q6, pregabalin 75mg BID. If refractory pain, tramadol 50mg q6 hours for breakthrough will be offered once taking PO, hydromorphone 0.2mg IV q2 as needed will be available if refractory pain and unable to take PO post operative day 0 (POD0). Regular diet will be allowed and encouraged on POD0. IV fluids will be given until POD1, and urine will be monitored q1 hour for the first 12 hours after which point the foley catheter will be removed. Subcutaneous heparin will be started POD1. Patients will also be given a bowel regimen consisting of docusate, senna glycoside and polyethylene glycol. If no bowel movement by POD1 and opioid use by patient, methylnaltrexone bromide will be administered. Patients will be encouraged to be out of bed (OOB) and ambulating as soon as possible POD0. Discharge criteria will be discussed and enforced with patient POD0.

Standard of care:

Preoperatively, patients will be randomly assigned to the standard of care. They will be instructed for clear liquid diet 24 hours prior to surgery with no food/liquid after midnight. On the day of surgery, they will receive subcutaneous heparin 5000 units as standard of care. They will have peripheral IV placed and be interview by the anesthesiology team in the preoperative holding area.

Intraoperatively, standard ASA monitors will be utilized and patients will receive general anesthesia with propofol, fentanyl, rocuronium (dosed by weight), and sevoflurane maintenance for all patients. Additional IV access will be established. Antibiotics will be administered within 1 hour of incision per protocol. Fluid management and hemodynamics will be treated as clinically indicated. All patients will receive ondansetron 4mg IV at the conclusion of the case for prevention of PONV.

Postoperatively, patients will return to PACU. Hydromorphone 0.2mg IV q30 minutes will be available for postoperative pain, and promethazine 6.25 mg IV BID or ondansetron 4mg IV q8 will be administered as needed for PONV. On return to the floor, IV fluids will be continued until patient is tolerating PO. Diet will be advanced per patient tolerance. IV hydromorphone 0.5mg q4 hours as needed will be available until patient is tolerating PO at which point oxycodone 5-10mg q4 as needed will be available for pain. Bowel regimen will be administered as needed, ambulation will be encouraged, and vital signs and urine output will be monitored per standard of care.

All patients will be discharged according to following criteria: independent ambulation, tolerating PO, baseline hemodynamics with urine output > 0.5 ml/kg/hr and adequate pain control with oral medications.

To assess the efficacy of the ERAS pathway, data collected will include postoperative pain scores and opioid use, time to first PO diet, time to return of bowel function, postoperative complications, incidence of PONV, and length of hospital stay. Patient satisfaction will be evaluated by the research team on the last day of hospitalization with a patient experience questionnaire (attached). Additionally, pain scores at follow-up appointments, additional hospitalizations and complications will be documented.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing this procedure who consent

Exclusion Criteria:

* patient refusal, female patients who are pregnant or nursing, patients with allergy to local anesthetic, American Society of Anesthesiology classification greater than 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-09-12 (Actual); Primary Completion 2023-06-12 (Estimated); Study Completion 2023-06-12 (Estimated)

PRIMARY OUTCOMES:
post operative opioid consumption | from time after discharge from PACU to discharge from the hospital (up to 7 days)
  amount of opioid pain medication required post operatively

SECONDARY OUTCOMES:
duration of hospitalization | from arrival on day of surgery to discharge from hospital (up to 7 days, anticipated 3 days)
  Hospital length of stay from day of surgery to discharge.
time to return of bowel function | arrival to PACU until discharge from hospital (up to 7 days)
  Post operative time to first sign of bowel function, either flatus or bowel movement.
time to first oral intake | from arrival to PACU until post-operative day 2 (48 hours)
  Post operative time following surgery until patient takes liquid/solid per os.
patient satisfaction | from discharge from PACU post operative day one to discharge home on last day of hospitalization (up to 7 days)
  Patient experience survey will be administered on last day of hospitalization. 14 question survery adapted from Cabellos M, et. al. Member of research team will distribute survey for completion by patients on last day of surgery. Survey focuses on pain management, communiation, recovery progression, facilities, and overall experience. Selection of open answer and likert scale questions.

CONTACTS AND LOCATIONS:
Overall Officials: Uzong Yoon, MD, MPH, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Background] Smith MD, McCall J, Plank L, Herbison GP, Soop M, Nygren J. Preoperative carbohydrate treatment for enhancing recovery after elective surgery. Cochrane Database Syst Rev. 2014 Aug 14;2014(8):CD009161. doi: 10.1002/14651858.CD009161.pub2. PMID 25121931
- [Background] Nemati E, Einollahi B, Lesan Pezeshki M, Porfarziani V, Fattahi MR. Does kidney transplantation with deceased or living donor affect graft survival? Nephrourol Mon. 2014 Jul 5;6(4):e12182. doi: 10.5812/numonthly.12182. eCollection 2014 Jul. PMID 25695017
- [Background] Rege A, Leraas H, Vikraman D, Ravindra K, Brennan T, Miller T, Thacker J, Sudan D. Could the Use of an Enhanced Recovery Protocol in Laparoscopic Donor Nephrectomy be an Incentive for Live Kidney Donation? Cureus. 2016 Nov 22;8(11):e889. doi: 10.7759/cureus.889. PMID 28018759
- [Background] McEvoy MD, Scott MJ, Gordon DB, Grant SA, Thacker JKM, Wu CL, Gan TJ, Mythen MG, Shaw AD, Miller TE; Perioperative Quality Initiative (POQI) I Workgroup. American Society for Enhanced Recovery (ASER) and Perioperative Quality Initiative (POQI) joint consensus statement on optimal analgesia within an enhanced recovery pathway for colorectal surgery: part 1-from the preoperative period to PACU. Perioper Med (Lond). 2017 Apr 13;6:8. doi: 10.1186/s13741-017-0064-5. eCollection 2017. PMID 28413629
- [Background] Meyer LA, Lasala J, Iniesta MD, Nick AM, Munsell MF, Shi Q, Wang XS, Cain KE, Lu KH, Ramirez PT. Effect of an Enhanced Recovery After Surgery Program on Opioid Use and Patient-Reported Outcomes. Obstet Gynecol. 2018 Aug;132(2):281-290. doi: 10.1097/AOG.0000000000002735. PMID 29995737
- [Background] Greco M, Capretti G, Beretta L, Gemma M, Pecorelli N, Braga M. Enhanced recovery program in colorectal surgery: a meta-analysis of randomized controlled trials. World J Surg. 2014 Jun;38(6):1531-41. doi: 10.1007/s00268-013-2416-8. PMID 24368573
- [Background] Ni X, Jia D, Chen Y, Wang L, Suo J. Is the Enhanced Recovery After Surgery (ERAS) Program Effective and Safe in Laparoscopic Colorectal Cancer Surgery? A Meta-Analysis of Randomized Controlled Trials. J Gastrointest Surg. 2019 Jul;23(7):1502-1512. doi: 10.1007/s11605-019-04170-8. Epub 2019 Mar 11. PMID 30859422
- [Background] Halawa A, Rowe S, Roberts F, Nathan C, Hassan A, Kumar A, Suvakov B, Edwards B, Gray C. A Better Journey for Patients, a Better Deal for the NHS: The Successful Implementation of an Enhanced Recovery Program After Renal Transplant Surgery. Exp Clin Transplant. 2018 Apr;16(2):127-132. doi: 10.6002/ect.2016.0304. Epub 2017 Aug 24. PMID 28836932